CLINICAL TRIAL: NCT03789526
Title: Ultrasound-guided Intervention and Hand Tenosynovitis in Patients With Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Abogamal, clinical professor of Rheumatology, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-AFMG 2018/6
Record Dates: First submitted 2018-12-24; First posted 2018-12-28 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Ultrasound Guided Injection
Keywords: Tenosynovitis; ultrasound; diabetes mellitus
MeSH Terms: conditions — Tenosynovitis; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: * Group one: 26 patients DM patients with tenosynovitis were injected by triamcinolone under ultrasound guidance.
  * Group two: 26 patients DM patients with tenosynovitis were injected by triamcinolone under clinical guidance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): * Group one: 26 patients DM patients with tenosynovitis were injected by triamcinolone under ultrasound guidance.
  Interventions: Procedure: ultrasound guidance
- Group 2 (No Intervention): Group two: 26 patients DM patients with tenosynovitis were injected by triamcinolone under clinical guidance.

INTERVENTIONS:
Procedure: ultrasound guidance — ultrasound guidance of tendon injection
  Arms: Group 1

SUMMARY:
Evaluates the efficacy of ultrasound guided versus clinically guided steroid injection in the management of tenosynovitis in DM patients.

DETAILED DESCRIPTION:
The current study will based on follow up study, conducted among patients presenting at outpatient rheumatology clinics of Al-Azhar University Hospitals, Egypt. with Diabetes mellitus duration at least 3 years and tenosynovitis of hand tendons with Richie tenderness grade 3.

All patients will randomized in two groups: Group one: 26 patients DM patients with tenosynovitis were injected by triamcinolone under ultrasound guidance. Group two: 26 patients DM patients with tenosynovitis were injected by triamcinolone under clinical guidance.

The affected tendons will scanned and scored for inflammation using ultrasound in all patients before the triamcinolone injection and then to be reassessed one month after the injection to determine the change in the tendons in both groups.

ELIGIBILITY:
Inclusion Criteria:

* • Diabetes mellitus.

  * Disease duration 3 years or more.
  * Tenosynovitis of hand tendons with Richie tenderness grade 3.

Exclusion Criteria:

* • Patients with recent hand trauma.

  * Patients with inflammatory hand arthritis.
  * Previous tendon surgery.
  * Previous tendon injection.
  * Patients with contraindication for injection as related infection, uncontrolled DM or bleeding tendency.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
change in Tenosynovitis pain | one month
  changes in VAS scale for pain,
change in Tenosynovitis tenderness | one month
  changes in Richie index for tenderness.
changes in ultrasound images of the Tenoasynovitis. | one month
  changes in Gery scale images, and power Doppler images of the tendons

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No